CLINICAL TRIAL: NCT01302353
Title: Phase I Trial of Emulsified Isoflurane in Adult Healthy Volunteers
Brief Title: Phase I Trial of Emulsified Isoflurane
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Dr. Jin Liu, Department of Anesthesiology, West China Hospital, Sichuan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PITEI; 2009L01628 (Other: State Food and Drug Administration of P.R. China)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Adverse Effect of Intravenous Anesthetics
Keywords: Phase I trial; Emulsified Isoflurane; Health volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- Arm 1 (0.0024 ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.0024ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 2 (0.006ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.006ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 3 (0.012ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.012ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 4 (0.02ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.02ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 5 (0.0301ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.0301ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 6 (0.0391ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.0391ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 7 (0.0508ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.0508ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 8 (0.066ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.066ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 9 (0.0859ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.0859ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 10 (0.1116ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.1116ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 11 (0.1451ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.1451ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 12 (0.1886ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.1886ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 13 (0.2452ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.2452ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 14 (0.3188ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.3188ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 15 (0.4144ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.4144ml/kg.
  Interventions: Drug: Emulsified Isoflurane
- Arm 16 (0.5387ml/kg) (Experimental): In this group, the volunteers receive emulsified isoflurane (120mg/ml) at the dose of 0.5387ml/kg.
  Interventions: Drug: Emulsified Isoflurane

INTERVENTIONS:
Drug: Emulsified Isoflurane

SUMMARY:
In this trial, our primary goal is to investigate the safety of intravenous infusion of emulsified isoflurane. In order to protect volunteers, the investigators adopt the modified Fibonacci dose-escalation, starting from a very low dose which is derived from the 1/600 of acute LD50 in pre-clinic study. The trial will be terminated if half of volunteers develop severe adverse event in any dose group or any volunteer develop fatal adverse event in any group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~45 years old (50:50 male:female) healthy volunteer;
* Body Mass Index (BMI) 19~24;
* health volunteers assessed by medical history and physical examination

  * systolic blood pressure between 100~140mmHg;
  * heart rate between 60~100bpm;
  * pulse oxygen saturation > 97% when inspiring air and reaching 100% after inspiring 100% oxygen for 5 min;
  * with normal result for routine lab test, including complete blood count, chemical test, urine test and stool test;
* Non-smoker and no history of alcohol or drug abuse;
* Fully understand the whole process of this trial and sign the informed consent.

Exclusion Criteria:

* Any history of allergy, especially to isoflurane or intralipid;
* Any suspected history of malignant hyperthermia in the volunteer or his/her relatives;
* Recent use of a medication with a pronounced effect on the central nervous system or any other organ (within 3 month)
* Recent participation in other clinical trial (within 1 month)
* Any history of difficult airway or suspected difficult airway;
* Pregnancy;
* Hyperlipidemia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Vital Signs | after drug infusion to 24 hours after infusion
  The vital signs include heart rate, cardiac rhythm, blood pressure, respiratory rate, pulse oxygen saturation, body temperature and end-tidal carbon dioxide.
  All the parameters are measured at the following time points:
  1. before drug infusion, recorded as baseline;
  2. every one minute, immediately from drug infusion to 15 min after infusion;
  3. every two minutes, from 15 min to 30 min after infusion;
  4. every five minutes, from 30 min to 60 min afeter infusion;
  5. every one hour, from 1 hour to 4 hours after infusion;
  6. 8 hours and 24 hours after infusion.

SECONDARY OUTCOMES:
Efficacy of emulsified isoflurane as an intravenous anesthetics | immediate from drug infusion, up to 24 hours after infusion
  This secondary outcome is an observational one only.
  The response to verbal command, to pain stimulus; and eyelash reflex are tested.
  The orientation and finger-to-nose test are also tested.
  The end-tidal partial pressure of isoflurane, observer's assessment of alertness/sedation (modified OAS/S score) and Bispectral index (BIS) are also recored.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, M.D, Principal Investigator — Department of Anesthesiology, West China Hospital, Sichuan University
Locations (1):
- Institute of Drug Clinical Trial• GCP Center,West China Hospital, Sichuan University, Chengdu, Sichuan, China